CLINICAL TRIAL: NCT00485940
Title: A Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of R108512 Tablets in Subjects With Chronic Constipation
Brief Title: Efficacy and Safety Study of Prucalopride for the Treatment of Patients With Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRU-USA-13
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Constipation
Keywords: constipation; prucalopride; QOL; SCBM; PAC-SYM
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Prucalopride 2 mg
  Interventions: Drug: Prucalopride
- 3 (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 2 (Active Comparator): Prucalopride 4 mg
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: Prucalopride — 2 mg o.d.
  Other Names: Resolor
  Arms: 1
Other: Placebo — Placebo o.d.
  Arms: 3
Drug: Prucalopride — 4 mg o.d.
  Other Names: Resolor
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether prucalopride is safe and effective in the treatment of chronic constipation

Hypothesis:

Prucalopride 2 mg and 4 mg given once daily for 12 weeks is superior to placebo for the treatment of patients with chronic constipation and is well tolerated in those patients

DETAILED DESCRIPTION:
This is a multicentre, Phase III trial with a parallel-group design, consisting of a 2 week drug-free run-in period, followed by a 12-week, double-blind, placebo-controlled treatment period.

During the run-in period, the subject's bowel habit will be documented and the existence of constipation confirmed. At the start of this period, all existing laxative medication will be withdrawn and subjects will be instructed not to change their diet or lifestyle during the trial. Subjects will be allowed to take a laxative (Dulcolax) as a rescue medication throughout the trial, but only if they have not had a bowel movement for three or more consecutive days. No Dulcolax or enemas should be taken within 48 hours prior to the start of double-blind treatment and 48 hours following the start of double-blind treatment. Subjects will enter the double-blind period if constipation is shown to be present during the run-in period.

If the definition of constipation is not met during the 2-week run-in, the subject will be considered ineligible for the double-blind period and will be discontinued from the study.

During the double-blind, randomised, placebo-controlled period, subjects will be treated for 12 weeks with either 2 mg or 4 mg R108512 or placebo, given once daily before breakfast.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant, non breast-feeding female outpatients at least 18 years of age (no upper age limit).
2. History of constipation; the subject reports, ona average,two of fewer spontaneous bowel movements per week that result in a feeling of complete evacuation and one or more of the following for at least 6 months before the selection visit:

   1. very hard (little balls) and/or hard stools at least a quarter of the stools
   2. sensation of incomplete evacuation following at least a quarter of the stools
   3. straining at defecation at least a quarter of the time. The above criteria are only applicable for spontaneous bowel movements, i.e., not preceded within a period of 24 hours by the intake of a laxative agent or by the use of an enema.

Subjects who never have spontaneous bowel movements are considered to be constipated and are eligible for the trial.

Exclusion Criteria:

1. Subjects in whom constipation is thought to be drug-induced, or subjects using any disallowed medication.
2. Subjects suffering from endocrine disorders, metabolic disorders or neurologic disorders.
3. Subjects with a megacolon/megarectum or a diagnosis of pseudo-obstruction.
4. Constipation as a result of surgery.
5. Known or suspected organic disorders of the large bowel, i.e. obstruction, carcinoma, or inflammatory bowel disease.
6. Subjects with severe and clinically uncontrolled cardiovascular, liver, or lung disease, neurologic or psychiatric disorders (including active alcohol or drug abuse), cancer or AIDS, and other gastrointestinal or endocrine disorders.
7. Subjects with impaired renal function.
8. Subjects with clinically significant abnormalities of haematology, urinalysis, or blood chemistry.
9. Females of child-bearing potential without adequate contraceptive protection during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 1998-03; Primary Completion 1999-05 (Actual); Study Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an average of 3 or more SCBM per week | 12 weeks

SECONDARY OUTCOMES:
Secondary efficacy variables: 1)Symptom variables 2)QOL variables | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John F Johanson, M.D., Principal Investigator — Private practice at Rockford Gastroenterology Associates Ltd. in Rockford

REFERENCES:
- [Result] Tack J, Stanghellini V, Dubois D, Joseph A, Vandeplassche L, Kerstens R. Effect of prucalopride on symptoms of chronic constipation. Neurogastroenterol Motil. 2014 Jan;26(1):21-7. doi: 10.1111/nmo.12217. Epub 2013 Sep 20. PMID 24106924
- [Derived] Lembo A, Staller K, Boules M, Feuerstadt P, Spalding W, Gabriel A, Youssef A, Xie Y, Terreri B, Cash BD. Efficacy and safety of prucalopride in patients with chronic idiopathic constipation stratified by age, body mass index, and renal function: a post hoc analysis of phase III and IV, randomized, placebo-controlled clinical studies. Therap Adv Gastroenterol. 2024 Dec 10;17:17562848241299731. doi: 10.1177/17562848241299731. eCollection 2024. PMID 39664231
- [Derived] Staller K, Hinson J, Kerstens R, Spalding W, Lembo A. Efficacy of Prucalopride for Chronic Idiopathic Constipation: An Analysis of Participants With Moderate to Very Severe Abdominal Bloating. Am J Gastroenterol. 2022 Jan 1;117(1):184-188. doi: 10.14309/ajg.0000000000001521. PMID 34585675
- [Derived] Tack J, Camilleri M, Dubois D, Vandeplassche L, Joseph A, Kerstens R. Association between health-related quality of life and symptoms in patients with chronic constipation: an integrated analysis of three phase 3 trials of prucalopride. Neurogastroenterol Motil. 2015 Mar;27(3):397-405. doi: 10.1111/nmo.12505. Epub 2015 Jan 11. PMID 25581251
- [Derived] Tack J, Quigley E, Camilleri M, Vandeplassche L, Kerstens R. Efficacy and safety of oral prucalopride in women with chronic constipation in whom laxatives have failed: an integrated analysis. United European Gastroenterol J. 2013 Feb;1(1):48-59. doi: 10.1177/2050640612474651. PMID 24917940